CLINICAL TRIAL: NCT05106088
Title: Variation in Humeral Head Bone Marrow Characteristics and Their Associations with Rotator Cuff Repair Healing
Brief Title: Variation in Humeral Head Bone Marrow Characteristics with Rotator Cuff Repair Healing
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kathleen Derwin, PhD, Associate Staff Scientist, The Cleveland Clinic
Other Study IDs: 21-811
Record Dates: First submitted 2021-10-14; First posted 2021-11-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Repairs
Keywords: longitudinal cohort, healing, imaging
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the time of rotator cuff repair, 8 ml of bone marrow will be aspirated from the humeral head for quantitative progenitor cell assays. A core biopsy at the tendon repair footprint will be collected for histologic analysis of bone marrow composition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study investigates correlations between humeral head bone marrow characteristics and tendon healing of rotator cuff repairs. The anticipated results would motivate future research aimed to investigate local enrichment or transplantation of connective tissue progenitor cells to augment rotator cuff repair and the pursuit of novel methods of bone marrow screening to preoperatively identify patients with bone marrow characteristics related to rotator cuff repair success or failure.

DETAILED DESCRIPTION:
Healing following rotator cuff repair (RCR) remains a significant clinical challenge, and repair failure rates of 20-30% continue to be reported. To date limited attention has been directed toward understanding how intrinsic mechanistic factors may contribute to variable healing rates following RCR. The objective of this proposal is to quantify the variability of the humeral head bone marrow in patients undergoing RCR and test the prognostic significance of the local concentration of connective tissue progenitors (CTPs) for tendon healing. Our approach will be to enroll 50 patients undergoing RCR. At the time of RCR, 8 ml of bone marrow will be aspirated from the humeral head for quantitative progenitor cell assays. A core biopsy at the tendon repair footprint will be collected for histologic analysis of bone marrow composition. Tendon healing will be assessed by MRI (Sugaya score) at 6 months follow-up, the timeframe in which majority of re-tears occur The variation of bone marrow characteristics among patients will be described (Aim 1) and their correlation with rotator cuff tendon healing will be investigated (Aim 2). The proposal seeks to shift the investigational paradigm to intrinsic patient biologic factors, a fundamental and under-investigated realm of potential prognostic factors of RCR healing. Demonstrating that humeral head characteristics associate with re-tear after RCR will support future work to develop tools to screen patient bone marrow for characteristics predictive of RCR success or failure and advance novel methods that promote local enrichment or transplantation of progenitor cells to augment RCR.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* 18-75 years
* 1-5 cm full thickness tear of the supraspinatus and/or infraspinatus tendon(s) that is fully reparable by double row technique as confirmed at surgery

Exclusion Criteria:

A 35 point exclusion criteria covers a variety of shoulder, musculoskeletal and general heath related conditions such as:

* prior shoulder surgery (including rotator cuff repair)
* symptomatic cervical spine disease
* a frozen shoulder-- defined as a loss of passive range of motion (ROM) of more than 20° in any plane compared to the contralateral shoulder
* advanced (grade 3 or 4) glenohumeral arthritis
* worker's compensation cases
* isolated subscapularis tears.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males or females, 18-75 years, with a 1-5 cm full thickness tear of the supraspinatus and/or infraspinatus tendon(s) requiring surgical repair
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Tendon healing | 6 months post-operation
  Sugaya score, 1-5 classification from MR imaging
Tendon healing | 6 months post-operation
  Tendon retraction (mm) from CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Derwin, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No